CLINICAL TRIAL: NCT04972851
Title: Autism Intervention Research Network on Behavioral Health: Self-Determined Learning Model of Instruction
Brief Title: AIRB-4: Self-Determined Learning Model of Instruction
Acronym: SDLMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of California, Davis (Other); University of Kansas (Other); University of Washington (Other); University of Pennsylvania (Other); University of Rochester (Other); Drexel University (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Human Development and Psychology, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-002001
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: autism; goals; school supports; determination
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNITED (Experimental): UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages within a few meetings and ongoing coaching from the research staff.
  Interventions: Behavioral: Self-Determined Learning Model of Instruction (SDLMI)
- Implementation as Usual (IAU) (Active Comparator): The organizations will implement SDLMI as usual. The research team will be available to provide support on the SDLMI intervention as needed.
  Interventions: Behavioral: Self-Determined Learning Model of Instruction (SDLMI)

INTERVENTIONS:
Behavioral: Self-Determined Learning Model of Instruction (SDLMI) — SDLMI is a teaching model that enables providers to teach students to:
  * make choices and decisions about setting a goal
  * develop action plans for academic or other goals
  * self-monitor and self-evaluate progress toward goal attainment
  * adjust the goal or plan

SUMMARY:
The AIRB research team will compare the use and effectiveness of each intervention (Mind the Gap, Remaking Recess and Self Determined Learning Model of Instruction) with and without the addition of our implementation strategy, UNITED. In all groups, the research team will train community practitioners using remote delivery of professional development modules specific to the intervention and active coaching as dictated by the intervention procedures.

The research team will pair UNITED with three interventions that cover the ages of early childhood, childhood, and adolescence. These include Mind the Gap (MTG), a family navigation intervention for children newly diagnosed under age 8, Remaking Recess (RR), a school-based social/peer engagement intervention for children ages 5-12, and Self-Determination Learning Model of Instruction (SDMLI), a self-advocacy intervention for adolescents (13-22 years; 22 is the upper age limit of high school for individuals with disabilities).

For the SDLMI, school personnel will be trained to work with adolescents with ASD using the SDLMI model. This model will help students with ASD set their own goals and help attain them. The total time commitment for the school personnel is 1 school year (2 semesters) for about 47 hours. The total time commitment for the parent of the student with ASD is about 1 hour (sign consent/fill out demographic survey). The total time commitment for the student with ASD is 1 school year (2 semesters) for about 25.25 hours.

DETAILED DESCRIPTION:
SDLMI targets school-based providers across grade levels (i.e., 6th - 12th grade) and disciplines (e.g., special education, general education). They will receive 7.5 hours of remote professional development in SDLMI. Coaching will take placed based on the SDLMI Facilitator Objectives that provide a road map for the facilitator. In school contexts, SDLMI instruction is implemented over the course of a school year or 2 semesters (approximately 24 weeks). Practitioners will receive 12 hours of remote coaching during sessions with students.

There will be 3 assessment time points. At entry, the teachers/school staff will fill out Demographic, Implementation Climate, Knowledge, Skills, and Use, and Acceptability of Intervention Measure (AIM). At 12 weeks of the study and at 24 weeks of the study (exit), they will fill out Implementation Climate, Knowledge, Skills, and Use, and Acceptability of Intervention Measure (AIM). Teachers/school staff will also fill out SDLMI fidelity questionnaire 6 times over the course of the school year. The parents will fill out a Demographic form at entry. Students will complete the following questionnaires at entry, mid-study (12 weeks) and end of study (24 weeks): the Self Determination Inventory: Student Report and Goal Attainment Scaling as a part of the SDLMI intervention.

All participants in SDLMI will be randomized to receive UNITED, exploratory implementation strategy, or implementation as usual (IAU). UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages. To address these requirements, the research team combined two well-tested strategies. The first is social network analysis (SNA) through which the research team will systematically identify members of the team who will implement each intervention. The second is TeamSTEPPS (Team Strategies and Tools to Enhance Performance and Patient Safety), an evidence-based set of teamwork tools that optimizes target population outcomes by improving communication and teamwork skills. The research staff will approach the school leaders (2 at maximum) and explain SDLMI. After the school leaders agree to participate in the study, they will complete a site agreement to participate and then fill out the Social Network Assessment (SNA) to provide names, roles, and emails of school personnel at the school that have significant roles in the school that relate to SDLMI. The research staff will then email these school personnel the SNA as well. After receiving the completed SNA assessments, the research staff will randomize each organization to UNITED vs Implementation as Usual (IAU). The research team will use the data from these assessments to assess both arms of the study. Additionally, for those randomized to UNITED, Dr. Elizabeth McGhee Hassrick at Drexel University and her team, will provide the research sites the top 2-5 school personnel identified by the SNA as key for intervention implementation support. This team will be invited to participate in the UNITED implementation team.

ELIGIBILITY:
Inclusion Criteria:

* school staff serving adolescents with ASD or NDD
* 63 adolescents ages 13-19 with ASD or NDD and family is under-resourced.
* Expert medical diagnosis or educational classification of ASD

Under-resourced, defined by:

* Attending a Title I school (a school that receives federal funding to improve the performance of economically disadvantaged students)or rural school
* Family income is under 250% of the federal guidelines for poverty rate (i.e., meets federal requirements to qualify for free or reduced lunch)
* Parent/Caregiver willing to participate

Exclusion Criteria:

* Personnel at school not working with adolescents with ASD or NDD
* Adolescents: under the age of 13 or over the age of 19, does not have ASD or NDD and family is not under-resourced.
* No official ASD/NDD diagnosis.
* Parent/Caregiver not willing to participate

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stages of Implementation Completion (SIC) | throughout study completion, an average of 18 months
  Tool developed by the Oregon Social Learning Center, is an 8 stage tool of implementation process and milestones, with stages spanning three implementation phases (pre-implementation, implementation, and sustainability.

SECONDARY OUTCOMES:
School Implementation Climate Scale | baseline,12 weeks, and 24 weeks
  This scale was adapted to be used by the research team to gather information from the schools/agencies in the study about the use of evidence-based practices in their organizations. It is rated from 0 to 4, with 0 being "not at all" and 4 being "very great extent." The higher the rating, the better the outcome.
Self-Determination Inventory (SDI-SR) | baseline, 12 weeks, and 24 weeks
  The Self-Determination Inventory (SDI) is comprised of a validated measure of self-determination created by researchers Karrie A. Shogren and Michael L. Wehmeyer at the University of Kansas. he SDI asks people to rate how they feel about their ability to be self-determined; that is to make choices, set and go after goals, and make decisions.
Goal Attainment Scaling (GAS) | baseline, 12 weeks, and 24 weeks
  The GAS is used to measure progress toward meeting goals. The goal is rated "much less than expected," "somewhat less than expected," "expected level of outcome," "somewhat more than expected," and "much more than expected." There is no numerical scaling, but a better outcome is expected from "much less" to "much more."
Social Network Survey | baseline, 12 months, and 18 months
  Survey created by the research team to gather information about the key people in each organization that can better support the SDLMI intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis MIND Institute, Davis, California
  - University of Kansas, Lawrence, Kansas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Locke J, Hassrick EM, Stahmer AC, Iadarola S, Boyd B, Mandell DS, Shih W, Hund L, Kasari C; AIR-B Network. Using Novel Implementation Tools for Evidence-based Intervention Delivery (UNITED) across public service systems for three evidence-based autism interventions in under-resourced communities: study protocol. BMC Psychiatry. 2022 Jul 16;22(1):478. doi: 10.1186/s12888-022-04105-9. PMID 35842614